CLINICAL TRIAL: NCT03357367
Title: Performance du TiVi Pour évaluer la réactivité Microcirculatoire de la Peau à l'Application d'un Courant Galvanique, Effet de l'Aspirine
Brief Title: TiVi Evaluation of Microcirculatory Reactivity of the Skin to Galvanic Stimulation: Effect of Aspirin
Acronym: PIRAAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A02528-45
Record Dates: First submitted 2017-11-20; First posted 2017-11-29 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAD patients (Experimental): Experimental: PAD patients Patients referred for vascular ultrasound investigation for suspicion of peripheral artery disease (PAD).
  Intervention is measurement of microvascular response to current application on the skin by TiVi system
  Interventions: Device: TiVi system

INTERVENTIONS:
Device: TiVi system — Device: TiVi system A galvanic current (0.1 mA) will be applied between 2 patches on the forearm of patient and protocol was repeated at 4 minutes.
  Microvascular response to current application (CIV) will be recorded by TiVi system 10 minutes later.
  Measurement of the value of skin blood flow (by TiVi system) at the stimulated area as compare to a non stimulated adjacent skin value taken as a reference Usual treatment will be recorded

SUMMARY:
Prospective interventional study. The aim is to analyze the effect of usual ongoing treatments over microvascular cutaneous response to galvanic current applications (CIV: current induced vasodilatation) with tissue vitality (TiVi) system on the forearm of subjects referred for ultrasound investigations due to suspicion of peripheral disease. Hypothesis is that the use of aspirin (even at low dose) abolishes the response.

This test could make it possible to detect the functional effects of low dose aspirin without using biological tests. A routine clinical application could be to use this CIV to verify adherence to aspirin.

DETAILED DESCRIPTION:
At admission eligible patients are proposed to participate. Written consent is signed after complete oral and written explanation of the protocol is signed.

No register of non-included patients will be kept. In included patients, in parallel to the routine ultrasound investigation for which the patient is referred, microvascular investigation will be performed as explained later in arm description.

Usual ongoing treatments are obtained by history and recorded. The end of the visit is the end of the participation of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* subjects referred for investigation of peripheral arterial disease.
* Affiliation to the French National healthcare system
* French speaking patients
* Ability to stand still for half a minute.

Exclusion Criteria:

* pregnancy
* inability to understand the study goal
* Patients protected by decision of law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2021-09-26 (Actual)

PRIMARY OUTCOMES:
Factor associated with CIV amplitude | 10 minutes after the second period of current application
  Determination of the coefficient r² characterizing the quality of the univariate linear regression explaining the Delta2 (maximum differential amplitude of the response to galvanic current between stimulated and non-stimulated zone) by the quantity of aspirin administered (expressed in mg).

SECONDARY OUTCOMES:
Role of aspirin in impaired CIV | 10 minutes after the second period of current application
  Likelihood ratio comparison of the univariate model to a multivariate model including all factors, primarily medicated, that may be associated with impaired CIV in vascular patients
Determination of the CIV cut-off value to optimally discriminate patients on aspirin from patients not taking aspirin | 10 minutes after the second period of current application
  Delta2 value (threshold CIV) minimizing distance to 100/100% sensitivity / specificity of receiver operating characteristics (ROC) analysis
Survival rate without major cardiovascular event (MACE) in patients with or without aspirin | at 12 months and 24 months
  the event-free survival rate is defined as the time between the inclusion date and the event date. If no event is observed at 24 months
Survival rate without major cardiovascular event (MACE)in patients with aspirin according to the CIV response. | at 12 months and 24 months.
  the event-free survival rate is defined as the time between the inclusion date and the event date. If no event is observed at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Samir MD HENNI, PhD, Principal Investigator — UH Angers
Locations (1):
- UH Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramondou P, Hersant J, Fouquet O, Sempore WY, Abraham P, Henni S. Current-Induced Vasodilation Specifically Detects, and Correlates With the Time Since, Last Aspirin Intake: An Interventional Study of 830 Patients. J Cardiovasc Pharmacol Ther. 2021 May;26(3):269-278. doi: 10.1177/1074248420971165. Epub 2020 Nov 7. PMID 33161777